CLINICAL TRIAL: NCT03521219
Title: Single Arm, Exploratory and Open Clinical Trial of Second-line Therapy With Apatinib Mesylate in Advanced Cholangiocarcinoma
Brief Title: A Study of Second-line Treatment With Apatinib for Advanced Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wei He, Deputy Chief Physician of Oncology, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP050
Record Dates: First submitted 2018-04-21; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): Apatinib 500mg, once a day, oral of each 28 day cycle. Number of cycle: until progression or unacceptable toxicity develops.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg, once a day, oral of each 28 day cycle. Number of cycle: until progression or unacceptable toxicity develops.

SUMMARY:
The propose of this study is to confirm safety and efficacy of Apatinib monotherapy in patients with advanced cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65 years;
2. Eastern Cooperative Oncology Group performance score (ECOG): 0-2;
3. Estimated survival time > 3 months;
4. Patients with recurrent or metastatic cholangiocarcinoma with histologic or cytological diagnosis;
5. Previous first-line GP programmes failed, or were not able to withstand first-line treatment;
6. At least one measurable lesion [spiral CT scan ≥ 10 mm (CT scan thickness not greater than 5mm)], Measurable lesions were not treated with radiotherapy or other topical treatments unless progress was achieved after treatment was completed (RECIST version 1.1);
7. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥ 1.5×109/L, PLT ≥ 75×109/L, HB ≥ 8 g/dL,ALB ≥2.8g/dL，TBIL ≤ 3×ULN, ALT or AST≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Cr clearance ≥ 50 mL/min;Thyroid function is normal；
8. No serious history of drug allergy；
9. Subjects volunteered for the study. Sign informed consent, good compliance, with follow-up.

Exclusion Criteria:

1. Patients have received targeted therapy；
2. Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, within 30 days after major surgery, uncontrolled high blood pressure medication, III-IV level cardiac insufficiency, severe liver and kidney dysfunction)；
3. Coagulation dysfunction (INR> 1.5, PT> ULN +4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment；
4. Urine routine showed that urine protein ≥++ or the urine protein in 24 hours>1.0 g；
5. Pregnant or lactating women；
6. History of other malignancy within 5 years except for effectively treated skin basal cell carcinoma, cutaneous squamous cell carcinoma and / or effectively excised orthotopic cervical and / or breast cancer;
7. The researchers judged other conditions that might affect clinical research and the outcome of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | 1 month
  the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease

SECONDARY OUTCOMES:
Progression-free Survival | 24 month
  Time from start of treatment until the first documented event of symptomatic progression or death.
Objective Response Rate(ORR) | 1 month, 3 month, 6 month
  Proportion of patients with reduction in tumor burden of a predefined amount
Overall Survival | 36 month
  from start of treatment to death from any cause, or last known date of survival

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China